CLINICAL TRIAL: NCT02063568
Title: The Use of Thromboelastometry (ROTEM) to Evaluate the Changes in Coagulation With Two Different Doses of Oxytocin Following Cesarean Delivery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Pro00051122
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-10

CONDITIONS: Coagulation Changes With Oxytocin
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Low dose oxytocin infusion (Active Comparator): oxytocin will be administered as an intravenous infusion at a rate of 0.33 units/min starting after fetal delivery upon umbilical cord clamping and continuing for a total of 30 minutes
  Interventions: Drug: Oxytocin
- High dose oxytocin infusion (Active Comparator): oxytocin will be administered as an intravenous infusion at a rate of 1.33 units/min starting after fetal delivery upon umbilical cord clamping and continuing for a total of 30 minutes
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin

SUMMARY:
The purpose of this study is to evaluate the differences in blood clotting seen in healthy patients given two different doses of oxytocin following cesarean delivery. The secondary objectives are to evaluate changes in blood pressure, rates of nausea and vomiting, and differences in blood loss with the two separate doses of oxytocin.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Age > or = 18 yrs
* Non-laboring women
* cesarean delivery under spinal anesthesia with pfannenstiel incision
* ASA I-III

Exclusion Criteria:

* Height <5'0"
* Allergy to phenylephrine
* Severe cardiac disease in pregnancy with marked functional limitations
* Women receiving NSAIDS, aspirin or other anticoagulants
* Subject enrollment in another study involving a study medication within 30 days of cesarean delivery
* Other physical or psychiatric condition which may impair the ability to cooperate with study data collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
coagulation as assessed by ROTEM | 30 minutes after oxytocin infusion started

SECONDARY OUTCOMES:
cardiac output changes with oxytocin | from start of surgery until 30 min after oxytocin infusion started
incidence of nausea and vomiting with oxytocin | from start of surgery until 30 minutes after oxytocin started
estimated blood loss with different doses of oxytocin | upon completion of surgery
changes in blood pressure with oxytocin | from start of surgery until 30 minutes after oxytocin started

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

REFERENCES:
- [Background] Solomon C, Collis RE, Collins PW. Haemostatic monitoring during postpartum haemorrhage and implications for management. Br J Anaesth. 2012 Dec;109(6):851-63. doi: 10.1093/bja/aes361. Epub 2012 Oct 16. PMID 23075633
- [Background] George RB, McKeen D, Chaplin AC, McLeod L. Up-down determination of the ED(90) of oxytocin infusions for the prevention of postpartum uterine atony in parturients undergoing Cesarean delivery. Can J Anaesth. 2010 Jun;57(6):578-82. doi: 10.1007/s12630-010-9297-1. Epub 2010 Mar 18. PMID 20238255
- [Background] Balki M, Erik-Soussi M, Kingdom J, Carvalho JC. Oxytocin pretreatment attenuates oxytocin-induced contractions in human myometrium in vitro. Anesthesiology. 2013 Sep;119(3):552-61. doi: 10.1097/ALN.0b013e318297d347. PMID 23676375
- [Background] Tita AT, Szychowski JM, Rouse DJ, Bean CM, Chapman V, Nothern A, Figueroa D, Quinn R, Andrews WW, Hauth JC. Higher-dose oxytocin and hemorrhage after vaginal delivery: a randomized controlled trial. Obstet Gynecol. 2012 Feb;119(2 Pt 1):293-300. doi: 10.1097/AOG.0b013e318242da74. PMID 22227638
- [Background] Butwick A, Harter S. An in vitro investigation of the coagulation effects of exogenous oxytocin using thromboelastography in healthy parturients. Anesth Analg. 2011 Aug;113(2):323-6. doi: 10.1213/ANE.0b013e3182222a82. Epub 2011 Jun 3. PMID 21642611
- [Background] Neuenschwander S, Pliska V. Effects of neurohypophyseal hormone analogues on blood clotting factor VIII and fibrinolytic activity in sheep. Eur J Pharmacol. 1997 Apr 4;323(2-3):205-13. doi: 10.1016/s0014-2999(97)00036-8. PMID 9128840